CLINICAL TRIAL: NCT01088750
Title: First International Inter-Group Study for Nodular Lymphocyte-Predominant Hodgkin's Lymphoma in Children and Adolescents
Brief Title: Surgery Alone or With CYC VBL and PRED or CVP Alone in Stage IA or IIA Nodular Lymphocyte-Predominant Hodgkin Lymphoma
Acronym: EuroNetLP1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Christine Mauz-Körholz (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); Euronet Worldwide (Other)
Responsible Party: Sponsor-Investigator, Christine Mauz-Körholz, Prof. Dr. Christine Mauz-Körholz, Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000667369; 2007-004092-19 (EudraCT Number)
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma
Keywords: childhood nodular lymphocyte predominant Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Cyclophosphamide; Prednisolone; prednylidene; Vinblastine; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery alone (Other): watch and wait strategy after complete resection of localised (e.g. Stage IA) nodular lymphocyte-predominant HL
  Interventions: Other: watchful waiting; Procedure: therapeutic conventional surgery
- CVP Chemotherapy (Experimental): 3 cycles of intensity-reduced, anthracycline-free chemotherapy (Cyclophosphamide, vinblastine and prednisone)
  Interventions: Drug: cyclophosphamide; Drug: prednisolone; Drug: vinblastine sulfate

INTERVENTIONS:
Drug: cyclophosphamide
  Other Names: CYC
  Arms: CVP Chemotherapy
Drug: prednisolone
  Other Names: PRED
  Arms: CVP Chemotherapy
Drug: vinblastine sulfate
  Other Names: VBL
  Arms: CVP Chemotherapy
Other: watchful waiting
  Arms: surgery alone
Procedure: therapeutic conventional surgery
  Arms: surgery alone

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, vinblastine, and prednisolone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Surgery to remove involved lymph nodes may be an effective treatment for young patients with nodular lymphocyte-predominant Hodgkin lymphoma.

PURPOSE: This phase IV trial is continuing to study the side effects of giving surgery alone or giving surgery with cyclophosphamide, vinblastine, and prednisolone compared with giving cyclophosphamide, vinblastine, and prednisolone alone in treating young patients with stage IA or stage IIA nodular lymphocyte-predominant Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 5-year event-free survival of children or adolescents with stage IA or IIA nodular lymphocyte-predominant Hodgkin lymphoma treated with surgery alone or with cyclophosphamide, vinblastine, and prednisolone.

Secondary

* Determine if this regimen results in a decrease in overall survival rates, in significant upstaging at relapse, or increased rates of histological transformation in these patients.

OUTLINE:

* Group 1 (patients with stage IA disease only): Patients undergo surgical resection of the involved lymph nodes. Patients who achieve complete resection then enter follow-up (watch and wait); patients who do not achieve complete resection enters group 2 treatment.
* Group 2 (patients with stage IIA disease or incompletely resected stage IA disease): Patients receive cyclophosphamide, vinblastine, and prednisolone for 3 courses. Patients with good response enter follow-up (watch and wait). Patients without a good response are taken off protocol.

After completion of study treatment, patients are followed-up periodically.

ELIGIBILITY:
Inclusion criteria:

* nodular lymphocyte-predominant Hodgkin's lymphoma confirmed by reference pathology.
* initial stage IA/IIA (according to local staging) or relapse stage IA or IIA and residual tumour after relapse biopsy and no additional surgery planned in nLP patients relapsing after surgery alone
* patient aged under 18 years at time of diagnosis
* written informed consent of the patient and/or the patient's parents or guardian according to national laws

Exclusion criteria

* pre-treatment of Hodgkin's lymphoma differing from study protocol
* Any extra-nodal involvement
* Inability to fulfil protocol requirements for imaging (CT, MRI, FDG-PET) at staging and response assessment
* known hypersensitivity or contraindication to study drugs
* prior chemotherapy or radiotherapy
* Current or recent therapy (within 30 days prior to the start of trial treatment) with steroids
* Current or recent (within 30 days prior to the start of trial treatment) treatment with another investigational drug or participation in another investigational trial
* other (simultaneous) malignancies
* severe concomitant diseases (e.g. immune deficiency syndrome)
* known HIV positivity
* pregnancy and / or lactation
* females who are sexually active refusing to use effective contraception (oral contraception, intrauterine devices, barrier method of contraception in conjunction with spermicidal jelly or surgical sterile) (except for surgery only)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 5 years
  Time from treatment start until relapse/progression, secondary malignancy or death

SECONDARY OUTCOMES:
Significant upstaging at relapse defined as development of B-symptoms, extranodal disease, or relapse higher than stage II | 5 years
  Stage greater than IIA at relapse diagnosis
Overall survival | 5 years
  Time from treatment start until death
Common Toxicity criteria toxicity Levels of therapy elements | 5 years
  Evaluation of AEs, SAEs atc. according to CTC
Complications of surgery | 5 years
  Listing of surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Koerholz, MD, Principal Investigator — Universitaetsklinikum Giessen und Marburg
Locations (1):
- Universitaetsklinikum Giessen-Marburg, Giessen, Germany

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/about-cancer/treatment/clinical-trials/search/v?a=8&id=NCI-2014-02026&loc=0&rl=2&st=C7258&t=C9357